CLINICAL TRIAL: NCT00428961
Title: Diabetic Genome Project: A Multi-Phase Prospective Registry to Identify Genetic Variation Among Diabetic Patients Undergoing Coronary Revascularization
Brief Title: Diabetes Genome Project: A Prospective Registry to Identify Genetic Variation Among Diabetic Patients
Acronym: DGP
Status: Completed | Type: Observational
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 03-102; ADA 7-04-CR-28
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Diabetes Mellitus; Insulin Resistance; Atherosclerosis
Keywords: diabetes mellitus; insulin resistance; atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood separated into 12 x1000µL, 10x500µL EDTA plasma, 2x1,000 µL and 20x200 µL of buffy coat (baseline only) and 2x1,000 µL of RBCs (baseline only)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Previous scientific research has found multiple genes that affect the risk for developing heart disease or complications during the treatment of heart disease. Less is currently known about how patients with heart disease may differ on the basis of other ailments they may have and how these other ailments may affect their treatment and prognosis. For this reason, researchers at the Mid America Heart Institute are conducting this research to find out how genes affect heart disease and recovery following angioplasty. The study will include patients with diabetes in order to determine if their genes are different from patients without diabetes.

A total of 1,607 patients were enrolled. There were 2 groups of patients selected for this study. The first group of patients included into the study will be those that are scheduled to have a diagnostic angiogram only. The second group of patients were those that had along with the angiogram a percutaneous transluminal coronary angioplasty, PTCA and or the use of a device called a coronary "stent", designed to help prop open the artery and to help avoid collapse. Samples for both groups will be stored for 30 years. After this time, all samples will be destroyed. Ultimately, we are hopeful that we will identify genes that will identify groups of patients at risk for heart disease.

DETAILED DESCRIPTION:
A single-center prospective registry which enrolled 1,607 patients. Following informed consent, patients underwent coronary angiography and/or percutaneous coronary intervention. This project was funded by an institution grant, philanthropy, industry, and a grant from the American Diabetes Association. The long-term goal is to better understand the biological underpinnings associated with diabetic atherosclerosis and vascular risk attributable to diabetes. All patients also provided informed consent for blood banking. Blood samples were collected at baseline (fasting) and in patients undergoing PCI (random) at 2,8 and 16 hours following arterial injury. These samples were separated in aliquots of 12 x1000µL, 10x500µL EDTA plasma, 2x1,000 µL and 20x200 µL of buffy coat (baseline only) and 2x1,000 µL of RBCs (baseline only). This protocol was designed to perform multiple biomarker studies as it avoids multiple freeze thaw cycles. A plaque imaging sub-study using the IVUS-VH software platform to characterize plaque tissue enrolled 209 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female gender
* Diabetes mellitus or no diabetes mellitus
* Candidate for percutaneous coronary intervention
* Informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Regional population attending a single-center specialty care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1607 (Actual)
Dates: Start 2002-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Marso, MD, Principal Investigator — University of Missouri Kansas City, Saint Luke's Hospital
Locations (1):
- Saint Luke's Hospital Mid America Heart Institute, Kansas City, Missouri, United States

REFERENCES:
- [Result] Marso SP, Mehta SK, Frutkin A, House JA, McCrary JR, Kulkarni KR. Low adiponectin levels are associated with atherogenic dyslipidemia and lipid-rich plaque in nondiabetic coronary arteries. Diabetes Care. 2008 May;31(5):989-94. doi: 10.2337/dc07-2024. Epub 2008 Feb 5. PMID 18252902
- [Derived] Lindsey JB, House JA, Kennedy KF, Marso SP. Diabetes duration is associated with increased thin-cap fibroatheroma detected by intravascular ultrasound with virtual histology. Circ Cardiovasc Interv. 2009 Dec;2(6):543-8. doi: 10.1161/CIRCINTERVENTIONS.109.876672. Epub 2009 Oct 13. PMID 20031772